CLINICAL TRIAL: NCT04117893
Title: Duloxetine Combined With Intra-articular Injection of Corticosteroid and Hyaluronic Acid Reduces Pain in the Treatment of Knee Osteoarthritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY 2019-086-02
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Osteoarthritis, Knee; Chronic Pain
Keywords: Osteoarthritis, Knee; Chronic Pain; hyaluronic acid; corticosteroid; duloxetine; Intra-articular injection
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain | interventions — Duloxetine Hydrochloride; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a prospective, randomized, open-label blind endpoint (PROBE) study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duloxetine combined with intra-articular injection (Experimental)
  Interventions: Drug: Duloxetine; Drug: intra-articular injection of corticosteroid and hyaluronic acid
- Intra-articular injection (Active Comparator)
  Interventions: Drug: intra-articular injection of corticosteroid and hyaluronic acid

INTERVENTIONS:
Drug: Duloxetine — Participants will start on duloxetine 30 mg per day for one week and then titrated up to duloxetine 60mg per day for 23 weeks.
  Arms: Duloxetine combined with intra-articular injection
Drug: intra-articular injection of corticosteroid and hyaluronic acid — Participants will receive a 3.5 ml intra-articular injection of 30mg of hyaluronic acid plus 10mg of triamcinolone acetonide.

SUMMARY:
Intra-articular injection of corticosteroid and hyaluronic acid is a common treatment for osteoarthritis of the knee. As a treatment drug for patients with depression, duloxetine has been shown in many studies to effectively relieve the pain of osteoarthritis and improve the function of the knee joint. However, there is no evidence regarding the efficacy of Intra-articular injection of corticosteroid and hyaluronic acid combined with duloxetine for pain management in patients with knee osteoarthritis. The aim of the study was to test the hypothesis that Intra-articular injection of corticosteroid plus hyaluronic acid combined with duloxetine could achieve superior pain management effects to Intra-articular injection of corticosteroid plus hyaluronic acid alone in patients undergoing knee osteoarthritis pain.

ELIGIBILITY:
Inclusion Criteria:

* Participants meet American College of Rheumatology clinical and radiographic criteria for the diagnosis of knee osteoarthritis with knee pain [ pain for ≥14 days of each month for ≥3 months before study entry, with a mean score ≥4 on the 24-h average pain score (0-10) using the average of daily ratings before the trial]
* Body mass index < 40 kg/m2
* Radiographic criteria included Kellgren-Lawrence grade Ⅱ-III
* Knee stability, no deformity, no lumbar spondylosis with radiculopathy.
* Good cognition, and the ability to understand the study protocol and the agreement to participate.

Exclusion Criteria:

* Inflammatory arthritis, autoimmune disorder, septic arthritis, or any other concomitant disease (such as liver and kidney disease)
* Those who prior synovial ﬂuid analysis indicative of a diagnosis other than osteoarthritis
* Participants with contraindications to duloxetine (currently using monoamine oxidase inhibitors, poorly controlled angle-closure glaucoma), previous exposure to duloxetine, combined with other drugs acting on the central nervous system (such as benzodiazepines) and allergic to any of the medications used in this study.
* With metabolic diseases or anticoagulation therapy
* Participants who had received invasive treatments to the knee during the past 6 months; joint replacement of the knee at any time or current infection in the affected limb.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Weekly mean of the 24h average pain scores | Twenty-fourth weeks
  Weekly mean of the 24h average pain scores in participants with osteoarthritis knee pain at the end of 24 weeks as reported in participants' diaries based on the 11-point Likert scale (an ordinal scale with 0 indicating 'no pain', and 10 indicating 'worst pain imaginable')

SECONDARY OUTCOMES:
The response to treatment | At weeks 1, 2, 4, 8, 16 and 24 post-injection
  The response to treatment defines as a 30% and a 50% reduction of weekly mean score in 24-h average pain severity ratings from baseline to endpoint at weeks1,2,4,8,16 and 24 post-injection.
The Brief Pain Inventory | At weeks 1, 2, 4, 8, 16 and 24 post-injection
  This is a self-reported scale that will use to measure the severity of pain and the interference of pain on function at weeks 1, 2, 4, 8, 16 and 24 post-injection. The severity of the pain was assessed by four questions: participants were rated on their most severe pain, their least severe pain, their average pain over the past 24 hours, and their current pain. The pain scale range from 0(no pain) to 10（extreme pain）. In the past 24 hours, seven questions assessed the impact of pain on daily activities, mood, walking ability, working normally, relationships with others, sleep and pleasure in life. The interference level ranges from 0(no interference) to 10(complete interference), and the average of the interference terms is obtained as a summary interference measurement.
The Western Ontario and McMaster Universities Osteoarthritis Index | At weeks 1, 2, 4, 8, 16 and 24 post-injection
  This instrument is designed to assess pain, stiffness, and physical function in participants with osteoarthritis of the knee and will be evaluate at weeks 1, 2, 4, 8, 16 and 24 post-injection. It consists of 24 questions: 5 on pain, 2 on stiffness, and 17 on physical function, each answered using a 5-point scale ranging from 0 (none) to 4 (extreme). Higher scores on the Western Ontario and McMaster Universities Osteoarthritis Index indicate worse pain, stiffness and functional limitations.
The Patient Global Impression of Improvement Scale | At weeks 2, 4, 8, 16 and 24 post-injection
  A patient-rated 7-point scale of symptomatic improvement, was assessed at all visits starting 2 weeks after treatment. On the The Patient Global Impression of Improvement Scale, a rating of 1 indicates that the participant is 'very much improved', a rating of 4 indicates that the participant has experienced 'no change', and a rating of 7 indicates that the participant is 'very much worse'. which range from 1 to 7.
Hospital Anxiety and Depression Scale | At weeks 2, 4, 8, 16 and 24 post-injection
  This self-rating patient-reported outcome measure will be developed to assess depression and anxiety in patients. Responses are rated on a 4-point Likert scale and range from 0 to 3, with higher scores indicating higher severity.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article will be shared after deidentification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The date will be shared from 6 months to 5 years following article publication.
Access Criteria: An independent review committee will be responsible for reviewing applications and purposes from investigators. The datasets used and/or analysed during the current study will be available from the corresponding author on reasonable request once the study has been completed.

REFERENCES:
- [Derived] Li DY, Han R, Zhao ZG, Luo F. Duloxetine combined with intra-articular injection versus intra-articular injection alone for pain relief in knee osteoarthritis: a study protocol for a randomised controlled trial. BMJ Open. 2020 Oct 27;10(10):e036447. doi: 10.1136/bmjopen-2019-036447. PMID 33109641